CLINICAL TRIAL: NCT03117920
Title: MinPAC: A Phase II, International Open Label Trial of Minnelide™ in Patients With Refractory Pancreatic Cancer.
Brief Title: A Phase II, International Open Label Trial of Minnelide™ in Patients With Refractory Pancreatic Cancer
Acronym: MinPAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Minneamrita Therapeutics LLC (Industry)
Collaborators: Barts & The London NHS Trust (Other); Translational Genomics Research Institute (Other); Stand Up To Cancer (Other); Cancer Research UK (Other); Lustgarten Foundation (Other); Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Minnelide002
Record Dates: First submitted 2017-03-16; First posted 2017-04-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Pancreatic Cancer
Keywords: Refractory pancreatic cancer; Minnelide; Minnelide002; 2017-000126-36
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 14-O-phosphonooxymethyltriptolide disodium salt

STUDY DESIGN:
Intervention Model Description: Single arm, open label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Minnelide (Experimental): 0.67 mg/m2 Minnelide daily as a 30min iv infusion on days 1-21 of each 28 day cycle, followed by a 7 day rest period (D 22-28).
  Interventions: Drug: Minnelide

INTERVENTIONS:
Drug: Minnelide — Minnelide will be administered at the dose of 0.67 mg/m2 as a 30 min infusion intravenously daily on days 1-21 of each cycle followed by a 7 day rest period (days 22-28).

SUMMARY:
MinPAC aims to see if the drug Minnelide can slow down tumour growth in patients with pancreatic cancer that is not responding to treatment. Minnelide is designed to rapidly release the anti-tumour molecule triptolide in the bloodstream and has been shown to slow cancer cell growth and induce cancer cell death. Minnelide is currently being investigated in other early phase trials and has shown promising response data.

There are strict eligibility criteria for this trial. Broadly speaking, patients with pancreatic cancer that has spread to other organs and has progressed on one or more chemotherapy regimens are eligible. Participants will receive Minnelide on days 1-21 of each 28 day cycle until their cancer stops responding to treatment. After that participants will be followed up 3 monthly for the collection of disease status and survival data.

MinPAC includes biological and imaging studies. Participants will be asked to donate tumour and blood samples and will be asked to undergo additional PET Scans. The study is being carried out in 4 sites in the UK and USA.

DETAILED DESCRIPTION:
MinPAC is an open label, international, multicentre phase II trial that aims to evaluate the effects of Minnelide treatment in patients with refractory pancreatic cancer. Eligible patients will receive Minnelide until disease progression unless there is evidence of unacceptable toxicity or the patient requests to be withdrawn from the study treatment. Once disease progression is documented, patients will enter a follow up phase during which data will be collected on further disease and survival status. If patients are unable to attend hospital visits during the follow up period then data will be collected either via telephone or via national registries with the patient's consent. The efficacy of Minnelide will be assessed on CT/MRI scan images and tumour and/or blood samples collected at baseline, during treatment and on completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Ability to comply with the protocol.
3. Aged ≥ 18 years.
4. Histologically or cytologically confirmed metastatic pancreatic adenocarcinoma that has progressed on one or more chemotherapy regimens.
5. Karnofsky performance status ≥ 70%.
6. At least one lesion that can be measured accurately at baseline as ≥10mm in the longest diameter (except lymph nodes which must have a short axis ≥15mm) with CT/MRI and which is suitable for repeated measurements per RECIST v1.1
7. Adequate haematological and end-organ function, as per the local institutions reference ranges, within 72 hrs prior to day 1 of cycle 1 of treatment defined by the following:
8. Life expectancy ≥ 12 weeks.
9. Negative pregnancy test within 14 days of day 1 cycle 1 for female patients of childbearing potential.
10. Tumour sites amenable to repeated biopsies.
11. Willingness to undergo paired tumour biopsies during the trial.
12. Agreement to use adequate contraception from 2 weeks before the start of treatment with Minnelide and until 90 days after completion of treatment.

Exclusion Criteria:

1. Patients with known or suspected brain metastasis
2. Significant cardiovascular disease such as New York Heart Associate Class III/IV, cardiac failure, myocardial infarction within 6 months prior to enrolment, unstable arrhythmia, or evidence of ischemia on ECG.
3. Baseline QTc exceeding 450msec (470msec for females) and / or patients receiving class 1A or class III anti-arrhythmic agents.
4. Known HIV, Hepatitis A, B or C infection.
5. Malignancies other than pancreatic cancer ≤5 years prior to Minnelide cycle 1 day 1, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcomes (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer or ductal carcinoma in situ treated surgically with curative intent) or localised prostate cancer treated with curative intent and absence of PSA relapse or incidental prostate cancer (Gleason score ≤3 +4 and PSA <10ng/L undergoing active surveillance and treatment naïve).
6. Severe infections ≤ 4 weeks prior to enrolment in the study as well as active, uncontrolled bacterial, viral or fungal infections requiring systemic treatment.
7. Major surgical procedure ≤ 2 weeks prior to enrolment or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis.
8. Treatment with chemotherapy or other investigational agents within 28 days (or at least 5 x the half-life of the drug) prior to day 1 cycle 1 of Minnelide™ (6 weeks for nitrosoureas or Mitomycin C).
9. Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational medicinal product (IMP) within ≤ 5 x the half-life of the IMP prior to day 1 cycle 1 of Minnelide.
10. Any other disease, metabolic dysfunction, physical examination finding or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of Minnelide, may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent.
11. Female patients who are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Disease Control rate (DCR) | Enrolment to 16 weeks
  DCR (CR+PR+SD) by RECIST v1.1

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Disease progression or death, assessed up to 18 months
  Time from enrolment until disease progression or death from any cause, whichever occurs first (RECIST v1.1)
Incidence of adverse events | Through completion of the safety visit an average of 4 months
  Adverse events by CTCAE v4.03
Overall survival (OS) | Death, assessed up to 18 months
  Time from enrolment until death
Response rate (RR) | Enrlolment to 16 weeks
  Percentage of individuals on study attaining a CR + PR (RECIST v1.1)
Change in tumour size and volume | Baseline to 8 weeks
  Change in the sum of diameters of the target lesions
Change in CA19-9 levels | Through completion of the treatment period an average of 4 months
  Percentage of patients with >20% decrease
Pharmacodynamic effect of Minnelide on tumour using PET Scans | 8 weeks
  Changes in SUV

OTHER OUTCOMES:
Biomarkers predictive of response to Minnelide | Through completion of the treatment period an average of 4 months
  Changes in circulating tumour stem cells.

CONTACTS AND LOCATIONS:
Overall Officials: David Propper, Principal Investigator — Barts & The London NHS Trust; Erkut Borazanci, Principal Investigator — HonorHealth Research Institute
Locations (3):
- United States (3):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Moores UC San Diego Cancer Center, La Jolla, California
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No